CLINICAL TRIAL: NCT05423093
Title: Pediatric Group Well Child Visits for Detection of Maternal Depression in Latinas
Brief Title: Virtual Group Psychoeducational Discussions With Spanish-Speaking Mothers of Infants in Pediatric Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00170216; 1K23MH118431-01A1 (NIH)
Record Dates: First submitted 2022-05-31; First posted 2022-06-21 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Postpartum Depression; Postpartum Anxiety
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention delivery (Experimental): Participants will receive a 45-60 minute single-session video group psychoeducational intervention delivered by clinic staff.
  Interventions: Behavioral: Single-Session Virtual Group Psychoeducational Session about Postpartum Depression

INTERVENTIONS:
Behavioral: Single-Session Virtual Group Psychoeducational Session about Postpartum Depression — Session contents include (1) Introduction to clinic staff, contacts, and resources (2) A video-recorded testimonial of a patient with a history of perinatal depression followed by a group discussion about/reflection on the video; (3) Review of prevalence and signs of PPD; (4) Discussion of clinic PPD screening procedures and rationale for screening; (5) Discussion of self-care and mood monitoring; (6) Discussion of relevant local resources, including information about availability of primary care resources for parents (including uninsured parents) and information about resources addressing social needs.

SUMMARY:
The goal of the proposed research is to test the feasibility and acceptability of a virtual group session which is intended to be offered universally to Spanish-speaking parents of newborns/infants attending pediatric primary care. The virtual session is intended to (1) enhance patient/family education about postpartum depression (PPD) and (2) Provide an orientation to families regarding relevant clinic and community psychosocial support resources available. The investigators will conduct a single-arm, open pilot of the session, which will be co-delivered by existing clinic staff (including social work and community outreach staff). Session contents include (1) Introduction to clinic staff, contacts, and resources (2) A video-recorded testimonial of a patient with a history of perinatal depression followed by a group discussion about/reflection on the video; (3) Review of prevalence and signs of PPD; (4) Discussion of clinic PPD screening procedures and rationale for screening; (5) Discussion of self-care and mood monitoring; (6) Discussion of relevant local resources, including information about availability of primary care resources for parents (including uninsured parents) and information about resources addressing social needs. The overall aim of the project is to Develop and pilot a virtual group augmentation of standard individual well-child care to improve (1) clinic screening procedures, discussion about and initial management of maternal depressive symptoms with immigrant Latinas and (2) patient symptom recognition, symptom disclosure, and subsequent treatment engagement

DETAILED DESCRIPTION:
The current study is designed as an open/single-arm pilot of the intervention (no comparison arm for this initial/preliminary study, which is also being offered as a clinic service).

Participants include Spanish-speaking parents of infants (6 months or younger) attending a pediatric practice.

Parents are recruited via flyers posted at the clinic as well as via referral from pediatric providers and staff (who can obtain permission from family for research staff to discuss the study with the family at the visit and/or to contact the family at a later time).

After screening, oral consent is obtained over the phone or zoom, and baseline measures are collected over the phone or zoom, prior to attendance at the intervention session.

Intervention Sessions will be offered at regular intervals, on at least a monthly basis, via Zoom. The sessions (desiged to last 45-60 minutes), which will be observed by research staff with permission of participants, are co-facilitated by a bilingual clinic social worker and bilingual community health worker.

Sessions consist of the following content:

1) Introduction and discussion of the purpose of the session/group; (2) Overview of services available at the clinic; (3) information about postpartum depression, including a five minute video testimonial followed by facilitated discussion about (a) prevalence and signs of postpartum depression, discussion of postpartum depression screening procedures and rationale for screening at the pediatric office, discussion of self-care and social support, and discussion of community resources (a list of resources are also mailed to the participants); (4) Discussion about insurance and health care for the infant and mother, including free/sliding scale clinics offering primary care for adults and rationale for engaging in one's own primary care in addition to pediatric health care for the infant.

After the session (within 2 weeks post-session) the research team collects post-session measures (see outcome measures) and conducts semi-structured interviews with participants.

6 months after the session, the research team will administer questionnaires over the phone assessing feedback about the intervention, physical and mental health services utilization, and post-intervention assessments (see outcome measures)

ELIGIBILITY:
Inclusion Criteria:

* Parent participants will be eligible if the preferred healthcare language is Spanish, if they are the mother of an infant (<2 months of age) attending participating pediatric practice, and if she is not felt to have a contraindication to participation (e.g., condition in the parent that would preclude the ability to reasonably participate in a virtual group session) by clinic staff
* Clinic staff participants - facilitators of virtual groups

Exclusion Criteria:

* <16 years old, preferred healthcare language not Spanish, not planning to attend participating practice, clinic staff determines contraindication to participation in group discussion

Ages: 16 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rheanna Platt, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fothergill KE, Gadomski A, Solomon BS, Olson AL, Gaffney CA, Dosreis S, Wissow LS. Assessing the impact of a web-based comprehensive somatic and mental health screening tool in pediatric primary care. Acad Pediatr. 2013 Jul-Aug;13(4):340-7. doi: 10.1016/j.acap.2013.04.005. PMID 23830020
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Eghaneyan BH, Killian MO, Sanchez K, Cabassa LJ. Psychometric Properties of Three Measures of Stigma Among Hispanics with Depression. J Immigr Minor Health. 2021 Oct;23(5):946-955. doi: 10.1007/s10903-021-01234-3. Epub 2021 Jun 19. PMID 34152503
- [Background] Caplan S. A Pilot Study of a Novel Method of Measuring Stigma about Depression Developed for Latinos in the Faith-Based Setting. Community Ment Health J. 2016 Aug;52(6):701-9. doi: 10.1007/s10597-016-0005-7. Epub 2016 Apr 16. PMID 27085546
- [Derived] Platt R, Richman R, Martin C, Martin KJ, Mendelson T. Feasibility and Acceptability of a Video Group Psychoeducational Intervention with Latina Immigrant Mothers to Enhance Infant Primary care. J Immigr Minor Health. 2024 Oct;26(5):945-952. doi: 10.1007/s10903-024-01612-7. Epub 2024 Jul 4. PMID 38963477
- See also: Rapid Risk Factor Surveillance System — https://www.rrfss.ca/questionnaires
- See also: National Latino and Asian American Study Documents — https://www.massgeneral.org/mongan-institute/centers/dru/research/past/nlaas-docs

RESULTS

PARTICIPANT FLOW:
Period: Consented Participants - Baseline Comple
Arm/Group | Intervention Delivery
Started | 26
Completed | 22
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Period: Attended Intervention Session
Arm/Group | Intervention Delivery
Started | 22
Completed | 19
Not Completed | 3
Not completed — Lost to Follow-up | 3
Period: Completed Post-intervention Measures
Arm/Group | Intervention Delivery
Started | 19
Completed | 16
Not Completed | 3
Not completed — Lost to Follow-up | 3
Period: 6-month Post Intervention Data Collected
Arm/Group | Intervention Delivery
Started | 16
Completed | 14
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: 26 participants consented, 22 were able to reached to complete baseline (pre-intervention) survey
Arm/Group | Intervention Delivery
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White, Hispanic | 9
  Race: Multiracial, Hispanic | 1
  Race: Black | 0
  Race: Other, Hispanic | 12
  Race: American Indian/Alaska Native | 0
  Race: Asian/Pacific Islander | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
Country of origin [Count of Participants; unit: Participants]
  El Salvador | 6
  Guatemala | 3
  Honduras | 6
  Ecuador | 2
  Mexico | 5
Maternal Education [Count of Participants; unit: Participants]
  8th grade or less | 14
  Some high school | 3
  High school or greater | 5
Time in United States [Mean (Standard Deviation); unit: years] | 11.5 (5.7)
Ever had mental health treatment [Count of Participants; unit: Participants]
  Yes | 6
  No | 16

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction as Assessed by the Intervention Satisfaction Survey
Description: Completed by parent participants. 5-point likert scale from 1 (strongly disagree) to 5 (strongly agree), higher scores indicative of higher satisfaction. No established cutoff.
Time Frame: Within 2 weeks of attending video group session
Population: Participants who completed the survey are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Delivery
Number analyzed (Participants) | 16
score on a scale | 4.06 (0.63)

2. Primary Outcome: Acceptability of Intervention Measure
Description: Completed by parent participants. 4-question pragmatic measure designed to assess construct of intervention acceptability as perceived by participant. 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree. Higher scores indicate greater acceptability. Score for each participant calculated as mean score for each item (range 1-5)
Time Frame: Within 2 weeks of attending video group session
Population: Participants who completed the survey are reported
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intervention Delivery
Number analyzed (Participants) | 16
units on a scale | 4.17 [4 to 5]

3. Secondary Outcome: Pre-Post Intervention Change in Mental Health Care Stigma as Assessed by the Stigma Concerns About Mental Health Care (SCMHC) Scale
Description: Completed by parent participants. The SCMHC is a 3-item measure assessing stigma-related barriers to the utilization of depression treatment (internalized stigma, fear of stigmatization, and stigma from family in seeking mental health care). Responses are coded as (0) disagree, (1) agree, and (7) don't know/refuse. Respondents receive one point for each response of "agree," which indicates agreement with the stigma-related barrier. The total scores range from 0 to 3 with higher scores indicating an increased internalization of stigma to mental health care
Time Frame: Baseline (pre-session); within 2 weeks post-session
Population: Participants who completed both pre and post-intervention survey are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Delivery
Number analyzed (Participants) | 16
score on a scale | -0.49 (0.97)

4. Secondary Outcome: Change in Depression Stigma as Assessed by the Adapted Personal Stigma Scale (PSS)
Description: 7 items, assess personal attitudes towards people with depression. Items answered on 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). Calculated as average item score, higher scores indicate higher levels of depression stigma.
Time Frame: Baseline (pre-session); within 2 weeks post-session
Population: Participants who completed both pre and post-intervention surveys are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Delivery
Number analyzed (Participants) | 16
score on a scale | -0.27 (0.31)

5. Secondary Outcome: Postpartum Depression Knowledge as Assessed by Adapted Postpartum Depression Knowledge Measure
Description: Measure of participant knowledge about postpartum depression knowledge- adapted and translated from the Ontario Rapid Risk Factor Surveillance Survey. Questions include whether the participant has heard of the concept of postpartum depression, asks participants to name symptoms of postpartum depression, and asks participants how common they would estimate the condition to be. There is no standard scale/scoring. Percent of participants answering affirmatively to the question "Have you heard of postpartum depression?" is reported.
Time Frame: Completed by participants at baseline (pre-session); within 2 weeks post-session; 6 months post session
Population: 22 participants completed this measure at baseline; 16 participants completed this measure 2 weeks post intervention; and 14 completed 6 months post intervention.
Measure: Number; unit: participants
Arm/Group | Intervention Delivery
Number analyzed (Participants) | 22
participants
  Yes - Baseline/Pre-session | 14
  No - Baseline/Pre-session | 8
  Yes - Within 2 weeks Post-session: number analyzed (Participants) | 16
  Yes - Within 2 weeks Post-session | 15
  No - Within 2 Weeks Post-session: number analyzed (Participants) | 16
  No - Within 2 Weeks Post-session | 1
  Yes - 6 Months Post-session: number analyzed (Participants) | 14
  Yes - 6 Months Post-session | 11
  No - 6 Months Post-session: number analyzed (Participants) | 14
  No - 6 Months Post-session | 3

6. Secondary Outcome: Intention to Disclose if Developed Postpartum Depression Symptoms as Assessed by Questionnaire
Description: Completed by parent participants. Single-question item: If I felt down, depressed, hopeless, or having little interest or pleasure in doing things I would try to contact someone at this clinic. Response options were No or Yes.
Time Frame: Baseline (pre-session); within 2 weeks post-session; and 6 months post-session
Population: 22 completed at baseline, 16 completed post-intervention, 14 completed at 6-month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Delivery
Number analyzed (Participants) | 22
Participants
  Pre-intervention: Yes | 22
  Pre-intervention: No | 0
  Post-Intervention: number analyzed (Participants) | 16
  Post-Intervention: Yes | 15
  Post-Intervention: No | 1
  6-month post intervention: number analyzed (Participants) | 14
  6-month post intervention: Yes | 14
  6-month post intervention: No | 0

7. Secondary Outcome: Intention to Seek Primary Care as Assessed by Survey Question
Description: Developed for this study, single likert scale question asked of participants who did not have an identified primary care doctor: As a result of the video group session, I plan to identify a doctor that I can see regularly for my own check-ups. Adapted from National Latino and Asian American Study. Scale range from 1-5, 1= strongly agree; 2=agree; 3=neutral/no opinion, 4=disagree, 5=strongly disagree
Time Frame: Baseline, Within 2 weeks of attending video group session, 6 months post intervention
Population: This question was only asked of participants who indicated not having a primary care provider at baseline, since it is about intention to identify/obtain a primary care provider in the future (so is not relevant to those who already have a primary care provider). Due to a technical error, the survey was inadvertently only administered to 6 of the 16 participants who completed 2 week post-intervention survey. It was administered to 14 participants 6-mo post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Delivery
Number analyzed (Participants) | 14
score on a scale
  Baseline | 2.71 (1.03)
  Post-intervention (within 2 weeks post intervention): number analyzed (Participants) | 6
  Post-intervention (within 2 weeks post intervention) | 1.83 (0.37)
  6-months post intervention | 2.07 (0.35)

8. Secondary Outcome: Self-reported Mental Health Service Utilization Within the Past 6 Months
Description: Single item, adapted from National Latino and Asian American Study; question: "within the past 6 months, have you had a therapy session with a psychologist or therapist or another professional that lasted 30 minutes or longer"?. Response options included "Yes", "No", "Unsure", and "Prefer Not to Answer".
Time Frame: 6 months post-intervention
Population: Participants who completed the 6-month post-intervention survey included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Delivery
Number analyzed (Participants) | 14
Participants
  Yes | 2
  No | 12
  Unsure | 0
  Prefer not to answer | 0

9. Secondary Outcome: Psychosocial Resource Utilization as Assessed by Questionnaire
Description: Completed by participant. Question developed for this project and translated/certified, assessing use of clinic ancillary services discussed in the intervention: In the past 2 months, have you used any of the resources that were discussed in the video session or on the clinic website? Responses could include "Yes", "No", or "Unsure"
Time Frame: 6-months post-intervention
Population: colleted from those who completed 6 month follow up survey (N=14)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Delivery
Number analyzed (Participants) | 14
Participants
  Yes | 4
  No | 9
  Unsure | 1

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Intervention Delivery
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT05423093/Prot_SAP_000.pdf